CLINICAL TRIAL: NCT01945411
Title: Assessment of Facial Measurements, the Length of Mouth Corner-mandible Angle and Incisors-mandible Angle, for Determining the Proper Sizes of Oropharyngeal Airway
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yonsei University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 4-2013-0440
Record Dates: First submitted 2013-09-04; First posted 2013-09-18 (Estimated); Last update posted 2015-07-31 (Estimated); Status verified 2015-07

CONDITIONS: General Anesthesia
Keywords: Airway Management; Ventilation
MeSH Terms: conditions — Respiratory Aspiration

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Experimental (Experimental): the length between incisor and mandible angle
  Interventions: Device: the length between incisor and mandible angle
- Active comparator (Active Comparator): the length between mouth corner-mandible angle
  Interventions: Device: the length between mouth corner-mandible angle

INTERVENTIONS:
Device: the length between incisor and mandible angle — the use of oropharyngeal airway (Guedel-type color coded oropharyngeal airway, Hudson RCI, Teleflex Medical, Research Triangle Park, NC) which size is the length between incisor and mandible angle
  Arms: Experimental
Device: the length between mouth corner-mandible angle — the use of oropharyngeal airway (Guedel-type color coded oropharyngeal airway, Hudson RCI, Teleflex Medical, Research Triangle Park, NC) of which size is the length between mouth corner and mandible angle
  Arms: Active comparator

SUMMARY:
The purpose of this study is to assess the facial measurements for determining the proper sizes of oropharyngeal airway. Investigators hypothesized that the length between incisors and mandible angle is more appropriate to estimate the size of oropharyngeal airway compared with the length between mouth corner and mandible angle.

ELIGIBILITY:
Inclusion Criteria:

* adult patients undergoing surgery that requires general anesthesia

Exclusion Criteria:

* anticipated difficult intubation
* patients without teeth or with loose teeth
* cervical spine disease
* upper airway disease
* body mass index over 35 kg/m2
* pregnancy

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 113 (Actual)
Dates: Start 2013-09; Primary Completion 2014-08 (Actual); Study Completion 2014-09 (Actual)

PRIMARY OUTCOMES:
proper size of oropharyngeal airway | up to 10 minutes after the start of anesthetic induction
  The oropharyngeal airway will be inserted into the patient's mouth. Investigators will check the laryngeal view using fiberoptic bronchoscope and the adequacy of ventilation after the investigator ventilates the patient using the mask. If both the laryngeal view and ventilation are appropriate, the size of oropharyngeal airway will be considered as the proper size for the patient.

CONTACTS AND LOCATIONS:
Locations (1):
- Severance Hospital, Seoul, South Korea

REFERENCES:
- [Derived] Kim HJ, Kim SH, Min NH, Park WK. Determination of the appropriate sizes of oropharyngeal airways in adults: correlation with external facial measurements: A randomised crossover study. Eur J Anaesthesiol. 2016 Dec;33(12):936-942. doi: 10.1097/EJA.0000000000000439. PMID 26908003